CLINICAL TRIAL: NCT02686970
Title: Spanish Adaptation and Study of Reliability of the European Quality Questionnaire (EuroQ2)
Status: Terminated | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Francisca Pérez-López, RN, Corporacion Parc Tauli
Other Study IDs: CorporationPT
Record Dates: First submitted 2016-01-18; First posted 2016-02-22 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2017-05

CONDITIONS: Critical Illness
Keywords: Family; Quality; Validate; ICU
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to adapt and validate to the Spanish the European Quality Questionnaire (EuroQ2) to evaluate families' experiences of quality of care for critically ill and dying patients in the ICU.

DETAILED DESCRIPTION:
The aim of this study is to adapt and validate a Spanish-language version of the European Quality Questionnaire (EuroQ2). Using a forward-backward translation methodology, we will translate the EuroQ2 into Spanish and will evaluate its psychometric characteristics in a clinical sample of 200 family members responsible for making medical decisions for patients who are discharged from the ICU or who died in the ICU. Cronbach's alpha values, confirmatory factor analysis (CFA) will be evaluated in order to know the reliability, construct validity, and convergent validity.

ELIGIBILITY:
Inclusion Criteria:

* Family members of patients admitted to the ICU for 48 hours or more.
* Family members responsible for patient decision making in the ICU who consent participate.

Exclusion Criteria:

* Family members younger than 18 years,
* Family members not able to read or write Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Family member or person responsible for patient decision making in the ICU
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
European Quality Questionnaire (euroq2) | 48 h after discharge of patients alive from ICU or 1 month after the death into ICU
  Opinions about Quality of care of ICU after the stay

CONTACTS AND LOCATIONS:
Overall Officials: Francisca Pérez-López, RN, MSc, Principal Investigator — Corporacion Parc Tauli
Locations (1):
- Corporacion Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jensen HI, Gerritsen RT, Koopmans M, Zijlstra JG, Curtis JR, Ording H. Families' experiences of intensive care unit quality of care: Development and validation of a European questionnaire (euroQ2). J Crit Care. 2015 Oct;30(5):884-90. doi: 10.1016/j.jcrc.2015.06.004. Epub 2015 Jun 16. PMID 26169545
- [Result] Gerritsen RT, Hofhuis JGM, Koopmans M, van der Woude M, Bormans L, Hovingh A, Spronk PE. Perception by family members and ICU staff of the quality of dying and death in the ICU: a prospective multicenter study in The Netherlands. Chest. 2013 Feb 1;143(2):357-363. doi: 10.1378/chest.12-0569. PMID 22878897